CLINICAL TRIAL: NCT07111351
Title: Multi-omics Studies of Primary Aldosteronism
Status: Recruiting | Type: Observational
Sponsor: Peking University First Hospital (Other)
Collaborators: Peking University (Other)
Responsible Party: Sponsor
Other Study IDs: 2025R0135
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-05

CONDITIONS: Primary Aldosteronism
MeSH Terms: conditions — Hyperaldosteronism | interventions — Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Aldosterone-producing adenoma
  Interventions: Other: Without intervention
- Idiopathic hyperaldosteronism
  Interventions: Other: Without intervention
- Primary Hpertension
  Interventions: Other: Without intervention
- Health control
  Interventions: Other: Without intervention

INTERVENTIONS:
Other: Without intervention — Without intervention

SUMMARY:
Primary aldosteronism is a prevalent yet underdiagnosed cause of secondary hypertension, contributing to significant cardiovascular morbidity and renal dysfunction. Despite affecting up to 20% of hypertensive patients, PA is frequently missed because it lacks distinctive clinical features and often presents with nonspecific symptoms like resistant hypertension or subtle electrolyte imbalances. The diagnostic pathway involves a stepwise approach: initial screening via the aldosterone-to-renin ratio, confirmatory testing (e.g., saline suppression or captopril challenge), and subtype differentiation using adrenal venous sampling to distinguish unilateral adenoma from bilateral hyperplasia. This complexity, combined with clinician unfamiliarity and variable access to specialized centers, perpetuates underdiagnosis. Early identification and tailored treatment are paramount in improving outcomes for patients with primary aldosteronism.

In this study, we will conduct a comprehensive multi-omics analysis on three sample types: 1) blood and urine samples from patients with primary aldosteronism, primary hypertension, and healthy controls; and 2) adrenal tissue samples from patients undergoing adrenalectomy for aldosterone-producing adenomas. We aim to systematically identify differentially expressed biomarkers that could serve as potential early diagnostic markers for primary aldosteronism. The findings may provide new insights into disease pathogenesis and contribute to improving early detection and personalized treatment strategies for this condition.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with primary aldosteronism , primary hypertension , or age- and sex-matched healthy controls;
2. Aged 18-80 years with complete medical records;
3. Willing to participate voluntarily and provide informed consent.

Exclusion Criteria:

1. History of chemotherapy or radiotherapy in the adrenal region ;
2. Positive serological or nucleic acid test results for HIV, hepatitis B, or hepatitis C , or a prior confirmed diagnosis;
3. Individuals with malignancies or autoimmune disorders ;
4. Study withdrawal during the trial period

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of participants recruited at Peking University First Hospital from May 2025 to May 2029. Eligible participants must meet all inclusion criteria: (1) diagnosis of primary aldosteronism, primary hypertension, or being age- and sex-matched healthy controls; (2) aged 18-80 years with complete medical records; and (3) voluntary participation with informed consent provision. Exclusion criteria include: (1) history of adrenal region chemotherapy/radiotherapy; (2) positive HIV/hepatitis B/C serology or prior diagnosis; (3) presence of malignancies or autoimmune disorders; and (4) withdrawal during the trial period. The study plans to enroll 400 patients.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2029-04-01 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Multi-omics data and analysis results | May 2025 to May 2029
  Collect various types of biological samples and utilize advanced proteomics and metabolomics technologies to obtain comprehensive omics data. Based on this, combine machine learning algorithms to deeply mine multi-omics data and clinical information, aiming to screen novel biomarkers for the prediction, classification, and diagnosis of primary aldosteronism, and construct a high-precision prediction model.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to ethical and practical considerations. The data contains sensitive personal health information, and sharing it could compromise participant confidentiality and privacy. Additionally, the study's institutional policies prioritize data security, limiting external access to protect against potential misuse or breaches. Ensuring compliance with ethical guidelines and institutional review board requirements further necessitates restricted data availability. While transparency in research is valued, these safeguards are essential to maintaining participant trust and adhering to data protection regulations.